CLINICAL TRIAL: NCT06197945
Title: Effects of Mulligan Bent Leg Raise With and Without Bowen Therapy on Hamstring Tightness in Asymptomatic Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0152
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Asymptomatic Condition
MeSH Terms: conditions — Asymptomatic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan bent leg raise (Experimental): The Mulligan Bent Leg Raise technique will be performed with 3 repetition, 3-4 times with 20 sec hold and one minute rest between each repetition.
  Interventions: Other: Mulligan bent leg raise
- Mulligan bent leg raise with Bowen therapy (Experimental): The Mulligan Bent Leg Raise technique will be performed with 3 repetition, 3-4 times with 20 sec hold and one minute rest between each repetition. After that Bowen therapy will be applied on hamstring bilateral.
  Interventions: Other: Mulligan bent leg raise with Bowen therapy

INTERVENTIONS:
Other: Mulligan bent leg raise — Mulligan bent leg raise
  Arms: Mulligan bent leg raise
Other: Mulligan bent leg raise with Bowen therapy — Mulligan bent leg raise with Bowen therapy
  Arms: Mulligan bent leg raise with Bowen therapy

SUMMARY:
Hamstring tightness is a common problem caused by a sedentary lifestyle and can have negative effects on posture and musculoskeletal function. It can lead to postural misalignment, increasing loading on the lumbar spine, increased pressure on inter-vertebral disc and potentially resulting in low back problems. Bowen technique and Mulligan Bent leg raise is used to treat conditions including hamstring tightness.

The goal of this clinical trial is to compare the effects of mulligan bent leg raise with and without Bowen therapy on hamstring tightness in asymptomatic adults.

DETAILED DESCRIPTION:
A randomized control trial will be conducted at Riphah Rehabilitation Center and Physiogic Physiotherapy clinic on 50 asymptomatic adults who meet the inclusion criteria will be recruited using non probability purposive sampling and randomly allocated using Random Allocation Software 2.0. Informed consent will be obtained from all participants. They will be divided into two groups which will contain 25 participants in each group. Group A will receive three alternate sessions of Mulligan Bent Leg Raise with Bowen therapy and Group B will receive three alternate sessions of Mulligan Bent leg Raise. The Mulligan Bent Leg Raise technique will be performed with 3 repetition, 3-4 times with 20 sec hold and one minute rest between each repetition.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* Age group between 18-40 years
* Unilateral limitation of SLR less than 75 degrees
* Asymptomatic, active knee extension less than 160 degrees

Exclusion Criteria:

* Fracture of Lower limb
* Individuals with soft tissue injury
* Chronic back pain
* Prolapsed Intervertebral disc
* Any surgery was done for back, pelvis hip or knee.
* Spinal deformity

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
Active Knee Extension Test | 1 week
  The Active Knee Extension Test is used to assess hamstring muscle length and the range of active knee extension in the position of hip flexion. A knee flexion angle of 20 ° or less is considered normal ROM on the AKE. The AKE has been found to have high reliability for intra-rater agreement (ICC = .86-.99) and moderate inter-rater reliability (ICC = .76-.89)
Sit and Reach Test | 1 week
  The Sit and reach test is one of the linear flexibility tests which helps to measure the extensibility of the hamstrings and lower back. Previous studies indicated that reliability estimate for Sit and reach test are consistently higher (.96 < R < .99)
Straight Leg Raise Test | 1 week
  also called the Lasegue test, Normal ROM for the PSLR has been reported as 80 ° of hip flexion. The PSLR has been reported to have high intra-rater (r = .91) and inter-rater (r = .93) reliability

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, Masters, Principal Investigator — Riphah International University
Locations (1):
- Physiogic Physiotherapy Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No